CLINICAL TRIAL: NCT00199992
Title: Platelets in Acute Wounds: A Pilot Study (PAWS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG-01-02-05
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Wounds
Keywords: acute wounds; wounds; platelets; platelet gel
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Procedure: application of autologous platelet gel

SUMMARY:
Comparison of wound healing treatments; platelet gel vs. control

DETAILED DESCRIPTION:
Comparison of autologous platelet gel to a control treatment in acute wounds, specifically punch biopsy wounds. Eight patients included in this pilot/feasibility study. Wound healing evaluated over 6 months for wound closure and long term outcome.

ELIGIBILITY:
Inclusion Criteria:

Healthy non-smokers, >18 years of age, BMI<30 -

Exclusion Criteria:

Smokers, obese, keloid formers, bleeding disorders, medications -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2005-01; Study Completion 2005-08

PRIMARY OUTCOMES:
Time to complete closure

SECONDARY OUTCOMES:
pain
long-term scar appearance

CONTACTS AND LOCATIONS:
Overall Officials: David HOM, M.D., Principal Investigator — Hennepin County Medical Center/ University of Minnesota
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Hom DB, Linzie BM, Huang TC. The healing effects of autologous platelet gel on acute human skin wounds. Arch Facial Plast Surg. 2007 May-Jun;9(3):174-83. doi: 10.1001/archfaci.9.3.174. PMID 17519207